CLINICAL TRIAL: NCT07321899
Title: Transcatheter Tricuspid Valve Replacement Using the Medtronic Intrepid™ TTVR System in Patients With Severe Symptomatic Tricuspid Regurgitation - PATHFINDER
Brief Title: Transcatheter Tricuspid Valve Replacement With the Medtronic Intrepid™ Transcatheter Tricuspid Valve Replacement (TTVR) System in Severe Tricuspid Regurgitation
Acronym: PATHFINDER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDT23032TMV006
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Severe Tricuspid Regurgitation
Keywords: Tricuspid Regurgitation; Symptomatic tricuspid regurgitation; Heart valve disease; Structural heart intervention; Severe valve disease; Randomized controlled trial; tricuspid insufficiency; tricuspid disease; tricuspid valve disease
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Medtronic Intrepid™ TTVR (Experimental): Transcatheter tricuspid valve replacement with Medtronic Intrepid™ TTVR System in patients with severe or greater tricuspid regurgitation.
  Interventions: Device: Medtronic Intrepid™ Transcatheter Tricuspid Valve Replacement (TTVR) System
- Edwards EVOQUE TTVR (Active Comparator): Transcatheter tricuspid valve replacement with Edwards EVOQUE TTVR in patients with severe or greater tricuspid regurgitation.
  Interventions: Device: Edwards EVOQUE Tricuspid Valve Replacement (TTVR) System
- Single Arm Registry (Experimental): Transcatheter tricuspid valve replacement with Medtronic Intrepid™ TTVR System in patients with severe or greater tricuspid regurgitation who are not eligible for randomization.
  Interventions: Device: Medtronic Intrepid™ Transcatheter Tricuspid Valve Replacement (TTVR) System

INTERVENTIONS:
Device: Medtronic Intrepid™ Transcatheter Tricuspid Valve Replacement (TTVR) System — Transcatheter Tricuspid Valve Replacement
  Arms: Medtronic Intrepid™ TTVR; Single Arm Registry
Device: Edwards EVOQUE Tricuspid Valve Replacement (TTVR) System — Transcatheter Tricuspid Valve Replacement
  Arms: Edwards EVOQUE TTVR

SUMMARY:
This clinical trial evaluates the safety and effectiveness of the Medtronic Intrepid™ Transcatheter Tricuspid Valve Replacement (TTVR) System in symptomatic patients with severe or greater tricuspid regurgitation.

DETAILED DESCRIPTION:
Prospective, global, pre-market, interventional, multi-center, randomized controlled pivotal trial to evaluate the safety and effectiveness of the Medtronic Intrepid™ Transcatheter Tricuspid Valve Replacement (TTVR) System compared to Edwards EVOQUE TTVR System in symptomatic patients with severe or greater tricuspid regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of consent.
* Severe symptomatic tricuspid regurgitation (TR) despite optimal medical therapy (OMT).
* Local site multidisciplinary heart team experienced in tricuspid valve therapies agrees that the subject is appropriate for TTVR.

Exclusion Criteria:

* Any tricuspid device currently in place.
* Anatomic contraindications.
* Need for emergent or urgent surgery.
* Left ventricular ejection fraction <25%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1186 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2031-09 (Estimated); Study Completion 2041-04 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Events (MAE) | 30-days post-procedure
Composite Endpoint: All-cause mortality, Heart failure hospitalization, and tricuspid valve reintervention | 1-year post-procedure

SECONDARY OUTCOMES:
Tricuspid regurgitation (TR) grade reduction | 6 months post-procedure
  Total number of patients with at least one grade TR reduction
Change in quality of life (QoL) as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline | 6 months post-procedure
  KCCQ overall summary score is a patient-reported measure of health status. Scores range from 0 to 100 where higher scores reflect better quality of life
All-cause mortality | 12 months post-procedure
Heart failure hospitalization | 12 months post-procedure
New onset conduction disturbance (NOCD) | 30 days post-procedure
Total procedure time | Procedure
Right ventricle (RV) dysfunction | 12 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Vinayak N. Bapat, MD, Principal Investigator — Minneapolis Heart Institute; Anita Asgar, MD, Principal Investigator — Northwestern Medicine Bluhm Cardiovascular Institute; Nicolas Dumonteil, MD, Principal Investigator — Clinique Pasteur Groupe CardioVasculaire Interventionnel; Azeem Latib, MD, Principal Investigator — Montefiore Medical Center; Firas Zahr, MD, Principal Investigator — Knight Cardiovascular Institute

IPD SHARING:
Plan to Share IPD: No